CLINICAL TRIAL: NCT03850743
Title: Biomarker Signatures of the Sleep-pain Enigma; a Collaborative Health Initiative Research Program (CHIRP) Funded Project
Brief Title: Biomarker Signatures of the Sleep-pain Enigma
Status: Completed | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Principal Investigator, Mary McDuffie, Research Nurse Manager, Defense and Veterans Center for Integrative Pain Management
Other Study IDs: 895846
Record Dates: First submitted 2018-12-10; First posted 2019-02-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2024-05

CONDITIONS: Post Surgical Pain and Sleep Impairment
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, prospective study that will leverage existing Standard of Care (SOC) patient reported outcomes (PRO) and Electronic Medical Record (EMR) data and collect additional Pain Rating Scale (PRS) data and blood samples from patients who consent to be in the study. Active duty service members and DEERS eligible patients who are injured and/or will undergo elective orthopaedic surgery are the target population.

DETAILED DESCRIPTION:
Sleep problems and pain, both acute and chronic, are common among military service members, reducing quality of life and military readiness. Evidence indicates sleep problems more strongly predict future acute and chronic pain than vice versa. This same pattern is also seen in the perioperative period, with sleep problems strongly predicting long-term post surgical pain. Though tightly linked, underlying biological mechanisms of the sleep-pain relationship in the perioperative period have yet to be identified, and treatment targets remain unknown. However, new technologies and methods in the areas of biomarker research (mRNA, microRNA, cytokine expression), as well as research describing psychosocial and clinical correlates, may help to identify patients most at-risk for long-term post-surgical sleep problems and pain, as well as identify new treatment targets.To address this research gap, the present observational study aims to collect four blood-samples from patients undergoing orthopedic surgeries at Walter Reed National Military Medical Center (WRNMMC) (N=240), both prior to and in the months following surgery, Additionally, patient reported outcomes, using the NIH's Patient Reported Outcome Measurement Information System (PROMIS), are collected as standard of care in the surgical clinics prior to surgery and for several years post-surgery. PROMIS scales cover a range of psychosocial (e.g., anxiety, depression, anger, social satisfaction, social isolation) and physical (e.g., fatigue, physical function) predictors. Through partnerships with the Defense and Veterans Center for Integrative Pain Management (USU), and WRNMMC Department of Orthopedic Surgery, the investigators will identify serum biomarkers (microRNA, cytokine expression) associated with pain and sleep-related outcomes prior to and in the months following surgery, as well as the role of psychosocial and clinical predictors, e.g. anxiety, depression, physical functioning, social functioning, opioid use) in outcomes. The long-term goal of this study are to understand risks for negative post-surgical outcomes, as well as help pave the way for future efforts to identify and test therapeutic interventions. Through this research, not only can the findings be used to improve surgical outcomes, but also increase quality of life among service members and force readiness.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military or DEERS eligible individuals
* Between the ages of 18 and 60 years old
* Able to understand written and spoken English
* Eligible for healthcare within Military Health Systems
* Having an orthopedic procedure at WRNMMC

Exclusion Criteria:

* Bleeding Disorder
* History of vasovagal response

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Active duty service members and DEERS eligible patients who are injured and/or will undergo elective orthopedic surgery. Up to 240 patients will be enrolled in this study at Walter Reed National Military Medical Center
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Biomarker Expression | Up to six months after surgery
  To determine the biomarkers (microRNA, mRNA, proinflammatory cytokines) associated with the presence (risk-related) or absence (resilience related) of sleep dysregulation and pain prior to surgery. To determine the biomarkers associated with increases/maintenance (risk-related) and decreases (resilience-related) of sleep dysregulation and pain chronification after surgery. Protein Biomarker Analysis: The cytokine expression analysis will be done using the Human Inflammatory Cytokines Multi-Analyte ELISArray Kit. The cytokines and chemokines to be tested with this array include IL1α, IL1β, IL2, IL4, IL6, IL8, IL10, IL12, IL17A, IFNγ, TNFα, and GM-CSF (Qiagen Inc.). For this analysis, we will use 50ul of serum samples along with the 50ul of assay buffer which will be loaded in the ELISA strips.

CONTACTS AND LOCATIONS:
Overall Officials: Chester C Buckenmaier, III, MD, Principal Investigator — Defense and Veterans Center for Integrative Pain Management
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03850743/ICF_000.pdf